CLINICAL TRIAL: NCT01341431
Title: Evaluation of the Symptomatic and Neuroprotective Effects of Bee Venom for the Treatment of Parkinson Disease
Brief Title: Bee Venom for the Treatment of Parkinson Disease
Acronym: MIREILLE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P090102
Record Dates: First submitted 2011-03-30; First posted 2011-04-25 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2013-06

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease; Bee venom; Motor fluctuations; Disease progression
MeSH Terms: conditions — Parkinson Disease; Disease Progression | interventions — Bee Venoms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- bee venom (Experimental)
  Interventions: Drug: bee venom
- saline (Placebo Comparator)
  Interventions: Drug: bee venom

INTERVENTIONS:
Drug: bee venom — 12 monthly injections of 100 micrograms(in 1 milliliter of NaCl 0.9%) of bee venom s.c.
  Other Names: 1: Experimental : Bee venom; 2: Placebo Comparator : NaCl 0.9%, 1 milliliter s.c.

SUMMARY:
The purpose of this study is to evaluate the efficacy of repeated (monthly) injections of bee venom on motor symptoms of Parkinson's disease over a period of one year, also the potential effects of this treatment on disease progression compared to placebo (saline injections).

DETAILED DESCRIPTION:
The investigators plan to assess the potential efficacy of repeated (monthly) injections of bee venom on the motor symptoms of Parkinson disease over a period of one year. The investigators will also assess the potential effects of this treatment on disease progression. All assessments will be conducted in comparison to placebo (saline injections).

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from Parkinson disease according to the Parkinson's Disease Society Brain Bank criteria (Hughes et al., 1992)
* Age > 40 ans (exclusion of juvenile forms)
* Hoehn and Yahr stage 1,5-3 off
* Pathological DaTSCAN
* MRI excluding atypical or secondary forms of parkinsonism
* Negative testing to bee venom (intradermoreaction)
* Affiliated to the French Social Security System

Exclusion Criteria:

* Parkinson disease Hoehn & Yahr stage < 1,5 or > 3
* Positive intradermoreaction to bee venom
* IgE positive to bee venom
* Known allergy to bee venom
* Contra-indications to treatment with bee venom (Alyostal®)
* Atypical or secondary parkinsonian syndrome (verified by MRI)
* Treatment with antipsychotics over the past 6 months
* Cardiac, hepatic or renal failure
* Normal DaTSCAN
* Contra-indications to MRI scanning
* Pregnancy
* Major depression or other severe acute/ongoing psychiatric disorder
* Cognitive impairment (MMS >24)
* Patient under guardianship

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
UPDRS III scores | one year
  Quantify the magnitude of a potential long-term symptomatic effect of bee venom by comparing UPDRS III scores at study inclusion and the final visit one year later before and after bee venom injection.

SECONDARY OUTCOMES:
Evaluate the potential effect of bee venom on disease progression by comparing UPDRS III off scores between treated/placebo group | one year
changes in L-Dopa equivalence doses over 12 months | 1 year
Correlate symptom (UPDRS III) progression with nigrostriatal denervation as measured by DaTSCAN | one year
Quantify the evolution (appearance, progression or regression) of motor fluctuations over the one year study period by UPDRS IV | > 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Hartmann, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Centre d'Investigation Clinique ICM, Paris, France

REFERENCES:
- [Derived] Hartmann A, Mullner J, Meier N, Hesekamp H, van Meerbeeck P, Habert MO, Kas A, Tanguy ML, Mazmanian M, Oya H, Abuaf N, Gaouar H, Salhi S, Charbonnier-Beaupel F, Fievet MH, Galanaud D, Arguillere S, Roze E, Degos B, Grabli D, Lacomblez L, Hubsch C, Vidailhet M, Bonnet AM, Corvol JC, Schupbach M. Bee Venom for the Treatment of Parkinson Disease - A Randomized Controlled Clinical Trial. PLoS One. 2016 Jul 12;11(7):e0158235. doi: 10.1371/journal.pone.0158235. eCollection 2016. PMID 27403743
- [Derived] Maurice N, Deltheil T, Melon C, Degos B, Mourre C, Amalric M, Kerkerian-Le Goff L. Bee Venom Alleviates Motor Deficits and Modulates the Transfer of Cortical Information through the Basal Ganglia in Rat Models of Parkinson's Disease. PLoS One. 2015 Nov 16;10(11):e0142838. doi: 10.1371/journal.pone.0142838. eCollection 2015. PMID 26571268